CLINICAL TRIAL: NCT07215858
Title: Randomized, Double-Blinded, Placebo-Controlled, Phase 2 Study of the Safety and Efficacy of BPL-1357 Against H1N1 Influenza Virus Challenge
Brief Title: BPL-1357 Against H1N1 Influenza Virus Challenge
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10002409; 002409-I
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10-16

CONDITIONS: Influenza; Human
Keywords: Influenza; Vaccine; Human Challenge
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): BPL-1357 given intramuscularly. Placebo given intranasally.
  Interventions: Biological: BPL-1357 IM; Other: Placebo IN
- Group B (Experimental): BPL-1357 given intranasally. Placebo given intramuscularly.
  Interventions: Biological: BPL-1357 IN; Other: Placebo IM
- Group C (Placebo Comparator): Placebo given intramuscularly and intranasally.
  Interventions: Other: Placebo IM; Other: Placebo IN

INTERVENTIONS:
Biological: BPL-1357 IM — Quadrivalent, inactivated, whole-virus vaccine containing 4 different wild-type avian viruses given intramuscularly.
  Arms: Group A
Biological: BPL-1357 IN — Quadrivalent, inactivated, whole-virus vaccine containing 4 different wild-type avian viruses given intranasally.
  Arms: Group B
Other: Placebo IM — Placebo given intramuscularly.
  Arms: Group B; Group C
Other: Placebo IN — Placebo given intranasally.
  Arms: Group A; Group C

SUMMARY:
Background:

Influenza (flu) infections are a serious global health threat. Each year, between 3 and 5 million people get the flu, and up to 500,000 die from it. Current vaccines protect against seasonal flus, but broader vaccines are needed to protect against potential flu pandemics.

Objective:

To test an experimental flu vaccine.

Eligibility:

Healthy people aged 18 to 55 years.

Design:

The study will last 5 to 8 months and has 2 phases, A and B.

The study vaccine will be given either as a shot in the arm or as a nasal spray. Participants will receive 1 of 3 combinations: (1) study vaccine in the nose and placebo in the arm; (2) placebo in the nose and study vaccine in the arm; or (3) placebo in the nose and placebo in the arm. A placebo is just like the real vaccine but contains no active ingredients.

Phase A: Participants will have 5 clinic visits over 56 days. They will receive a shot and a nasal spray at 2 of the visits, 28 days apart. At each visit, they will have a physical exam, with tests of their blood, urine, and nasal secretions. They will check their temperature at home and record any symptoms for 7 days after each vaccine.

Phase B: Participants will stay in the hospital for at least 9 days. They will be infected with a flu virus. They will provide blood, urine, and nasal fluid samples. They will have tests of their heart function. They will remain in the hospital until they test negative for the flu 2 days in a row.

They will have 2 follow-up visits, 4 and 8 weeks after leaving the hospital.

DETAILED DESCRIPTION:
Study Description:

This is a randomized, double-blinded, placebo-controlled, multicenter, phase 2 clinical trial of beta-propiolactone (BPL)-inactivated quadruple influenza virus cocktail vaccine (BPL-1357) administered intramuscularly (IM) or intranasally (IN) in 2 doses 28 days apart. The study has 2 phases: a vaccination phase (Phase A) and a challenge phase (Phase B). In phase A participants will be randomized to 1 of 3 groups for treatment assignment: group A IM BPL-1357 plus IN placebo, group B IM placebo plus IN BPL-1357, or group C IM placebo and IN placebo. In phase B, participants will undergo influenza challenge as inpatients. The primary hypothesis is that IN and IM BPL-1357 will be safe and offer protection against mild-moderate influenza disease (MMID) caused by H1N1 influenza challenge compared to placebo.

Objectives:

Primary Objective:

1. To measure the efficacy of BPL-1357, given IM or IN, in preventing MMID compared to placebo.
2. To assess the safety of BPL-1357, given IM or IN as 2 doses 28 days apart, including after H1N1 influenza challenge.

Secondary Objective:

1. To assess the correlates of protection associated with BPL- 1357 against H1N1 influenza challenge.
2. To measure the efficacy of BPL-1357, given IM or IN, in reducing total InFLUenza Patient Reported Outcome (FLUPRO) scores compared to placebo.
3. To measure the efficacy of BPL-1357, given IM or IN, in preventing shedding measured by quantitative real-time polymerase chain reaction (rtPCR) compared to placebo.
4. To measure the efficacy of BPL-1357, given IM or IN, in reducing shedding duration measured by rtPCR compared to placebo.
5. To assess the immunogenicity of BPL-1357 given IM or IN.

Tertiary Objective:

1. To characterize the systemic and mucosal humoral immune responses induced by BPL-1357 at multiple timepoints before and after influenza challenge.
2. To further characterize the immune response induced by BPL-1357 and subsequent influenza challenge through variable, diversity, and joining (VDJ) gene repertoire analysis, cytokine analysis, cytometry, transcriptomics, and further assessment of B- and T-cell responses.
3. To assess time-from-vaccination with clinical outcomes.
4. To assess HLA types with immune responses.
5. To assess BPL-1357 vaccine efficacy against any community-acquired influenza during the study.

Endpoints:

Primary Endpoints:

1. Efficacy: Rate of MMID, defined as a positive US Food and Drug Administration (FDA) - approved clinical test for influenza plus 1 or more influenza symptoms.
2. Safety:

   1. Solicited adverse events (AEs) occurring within 7 days of each vaccination dose recorded through questionnaires.
   2. Unsolicited AEs occurring within 28 days of each vaccination dose.
   3. Serious adverse events (SAEs) occurring through study completion or withdrawal from study.

Secondary Endpoints:

1. Correlations and relationships between clinical outcomes and immune responses.
2. Total FLU-PRO questionnaire scores after influenza challenge.
3. Proportion of patients who shed virus after influenza challenge as measured by rtPCR.
4. Mean duration (days) of shedding as measured by rtPCR.
5. Immunogenicity at 28 days after vaccine dose 2 (PAD56):

   1. Antibodies against H1, H3, H5, and H7 head and stalk as measured by hemagglutination inhibition (HAI) or enzyme-linked immunosorbent assay (ELISA) from blood and mucosal samples at PAD56.
   2. Antibodies against N1, N3, N8, and N9 as measured by neuraminidase inhibition (NAI) or ELISA from blood and mucosal samples at PAD56.

Tertiary Endpoints:

1. Additional antibody titer characterization via:

   1. Antibodies against H1, H3, H5, and H7 head and stalk as measured by HAI or ELISA from blood and mucosal samples at all timepoints.
   2. Antibodies against N1, N3, N8, and N9 as measured by NAI or ELISA from blood and mucosal samples at all timepoints.
2. Additional immune response characterization through:

   1. VDJ gene repertoire analysis.
   2. Cytokine analysis.
   3. Flow cytometric phenotyping of lymphocytes.
   4. Transcriptomic gene expression.
   5. B- and T-cell responses.
3. Correlations and relationships between time-from-vaccination and clinical outcomes and immune responses.
4. Relationship between HLA types and immune responses.
5. Integrated challenge endpoints (e.g., MMID, infection) with any community acquired influenza diagnosed while on study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

1. Adults >=18 and <= 55 years of age at the time of consent.
2. Able to provide written informed consent.
3. Non-smoker (i.e., tobacco and cannabis) and does not use vape or e-cigarette products currently. Also, must not have used any of these products extensively in the past (regular use more than 5 times per week, more than 6 months lifetime total).
4. Has not received influenza vaccination of any type within 8 weeks (about 2 months) prior to enrollment and consents to not receive influenza vaccination of any type until after the end of study participation (PBD63).
5. Has not received any other vaccination of any type within 4 weeks prior to enrollment and consents to not receive any unlicensed vaccine until after the end of the study (PBD63).
6. Has not received any broadly protective influenza vaccine in the past.
7. Participants of childbearing potential must meet one of the following criteria through the end of study participation (PBD63):

   1. Is infertile, including postmenopausal status (as defined by age .45 years plus no menses for >= 1 year without an alternative medical cause) or history of hysterectomy or bilateral oophorectomy.
   2. Agrees that, when engaging in intercourse that can result in pregnancy, they will use an acceptable or highly effective form of contraception, and their male partner will use a condom with spermicide. Acceptable methods of female contraception include

   the following:
   * Bilateral tubal ligation
   * Implant of levonorgestrel
   * Injectable progestogen
   * Oral contraceptive pills
   * Diaphragm with spermicide
   * Intrauterine device (IUD)
   * Sexual abstinence
   * Vasectomized partner
8. Able to speak and understand English (NIH).
9. Able to speak and understand English and/or Spanish (UTMB).
10. A negative HIV test within 6 months before enrollment.
11. Has not used IN medications (including but not limited to nasal sprays, sinus rinses), and has not routinely used over-the-counter medications (including but not limited to aspirin, decongestants, antihistamines, and other nonsteroidal anti-inflammatory drugs), and herbal medications (including but not limited to herbal tea or St. John fs Wort) within 14 days (about 2 weeks) prior to study enrollment and agrees not to use these medications until after the end of study participation (PBD63), unless approved by the investigator.
12. Agrees not to donate blood or blood products from enrollment through the final study visit (PBD63).
13. Not planning on cohabitating with any high-risk individuals (e.g., infants, elderly, those with high-risk conditions (e.g., pregnancy, medical conditions such as those outlined in exclusion criterion 1) for at least 2 weeks after discharge from the inpatient portion of this study.
14. Participant is willing and able to comply with all trial procedures.

EXCLUSION CRITERIA

Individuals meeting any of the following criteria will be excluded from study participation:

1. Current medical conditions (self-reported or medically documented) including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression, immune deficiency, or ongoing malignancy.
   5. Neurological and neurodevelopmental condition (e.g., Bell s palsy, cerebral palsy, epilepsy, seizures).
2. Body mass index (BMI) <18 and >35.
3. Pregnant or breastfeeding.
4. History of postinfectious or postvaccine neurological sequelae including GBS.
5. History of stroke within the past 5 years.
6. Acute illness within 7 days prior to enrollment (PAD0).
7. Known allergy to influenza vaccination or components contained in the influenza vaccine being used.
8. Known allergy to influenza treatments (including oseltamivir or nonsteroidal anti-inflammatory medications).
9. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
10. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
11. Receipt of any unlicensed drug or investigational agent within 3 months or 5.5 half-life (whichever is greater) prior to enrollment.
12. Receipt of any unlicensed vaccine within 6 months prior to enrollment.
13. Self-reported or known history of alcoholism or drug abuse or use within 6 months prior to enrollment, or positive urine test for illicit drugs (i.e., amphetamines, cocaine metabolites, benzodiazepines, opiates, but not tetrahydrocannabinol) prior to vaccination on PAD0.
14. Self-reported or known history of psychiatric or psychological issues that require treatment and are deemed by the PI to be a contraindication to protocol participation.
15. History of angioedema or anaphylaxis.
16. Study site staff who directly report to the study or site PI are excluded from participation.
17. Any condition, event or lab value that, in the judgment of the investigator, is a contraindication to protocol participation or would place the participant at increased risk for participation.
18. Any condition or event that, in the judgment of the investigator, impairs the participant's ability to give informed consent.

Individuals meeting any of the following criteria will be excluded from participation in Phase B:

1. Positive urine test for illicit drugs (i.e., amphetamines, cocaine metabolites, benzodiazepines, opiates, but not tetrahydrocannabinol) prior to inoculation (PBD0).
2. Acute illness within 7 days prior to inoculation with the human challenge virus (PBD0).
3. Grade 3 or greater sign, symptom, or lab abnormality that is clinically significant and (in the opinion of the site PI) puts the participant at higher risk of adverse effects with influenza challenge.
4. Pregnant or breastfeeding.
5. Positive test for influenza within 8 weeks prior to challenge.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety (solicited AEs 7 days after vaccination, unsolicited adverse events (AEs) within 28 days post-vaccination, serious AEs (SAEs) | 15-25 weeks
  Safety of the vaccine will be assessed, including standardized measurement of immediate reactogenicity by symptom survey, as well as long-term follow-up for any SAEs, including after challenge, will be performed.
Rate of mild-to-moderate influenza disease (MMID), defined as a positive US FDA-approved clinical test for influenza plus one or more influenza symptoms | 7-17 weeks
  Rate of MMID will be compared across groups to estimate vaccine efficacy.

SECONDARY OUTCOMES:
Immunogenicity at 28 days after vaccine dose 2 (PAD56): | 8 weeks
  Antibodies against N1, N3, N8, and N9 and H1, H3, H5, H7 head and stalk as measured by NAI, HAI and/or ELISA from blood and mucosal samples to assess immunogenicity.
Mean duration (days) of shedding as measured by rtPCR. | 7-17 weeks
  Vaccine, IM or IN, may affect the duration of shedding.
Proportion of patients who shed virus after influenza challenge as measured by rtPCR. | 7-17 weeks
  Vaccine, IM or IN, may affect the rate of infection (whether symptomatic or asymptomatic).
Total FLU-PRO questionnaire scores after influenza challenge. | 7-17 weeks
  Vaccine, IM or IN, may affect duration and severity of symptoms as measured by FLU-PRO, a validated survey tool for measuring severity of symptoms with influenza.
Correlations and relationships between clinical outcomes and immune responses. | 7-17 weeks
  Post-vaccine measurements of immune response will be correlated with clinical outcomes to understand mechanisms of vaccine protection.

CONTACTS AND LOCATIONS:
Overall Officials: Luca T Giurgea, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Texas Medical Branch, Galveston, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002409-I.html